CLINICAL TRIAL: NCT00886587
Title: A Double-Blind, Randomized, Active-Controlled Clinical Trial To Evaluate the Safety and Efficacy of a New Device in the Management of Mild to Moderate Atopic Dermatitis in Children
Brief Title: To Evaluate the Safety and Efficacy of a New Device in the Management of Mild to Moderate Atopic Dermatitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EMOECZ0002
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Atopic Dermatitis
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 11054-010 (Experimental): F# 11054-010 Investigational Device
  Interventions: Device: F# 11054-010
- 10495-053 (Active Comparator): F# 10495-053 Atopiclair
  Interventions: Device: F# 10495-053

INTERVENTIONS:
Device: F# 11054-010 — Apply 3 times daily (or as needed) on all body areas, including the affected areas of the body and face throughout duration of study. Massage gently into skin.
  Other Names: Investigational Device
  Arms: 11054-010
Device: F# 10495-053 — Apply 3 times daily (or as needed) on all body areas, including the affected areas of the body and face throughout duration of study. Massage gently into skin.
  Other Names: Atopiclair® Skin and Wound Emulsion
  Arms: 10495-053

SUMMARY:
The purpose of this study was to evaluate the safety of the investigational study product and see how well it works to relieve signs and symptoms of children with mild to moderate Atopic Dermatitis (AD), also known as eczema, in comparison to that of a similar marketed product. This study was conducted to assess the safety of the investigational new study product and how well it works to treat AD in children, by making AD visually better, and reducing the amount of itch.

DETAILED DESCRIPTION:
This was a multi-center, double-blind, randomized, active-controlled trial in children 2 to 12 years of age with mild to moderate AD. A sufficient number of subjects were screened to ensure that approximately 80 subjects were randomized, to yield 70 completed subjects. Subjects were randomized to one of the two treatment groups: the J&J Device or Atopiclair®. All subjects were to return to the clinical site for clinical assessments at baseline (Day 1) and at Days 3, 8, 15, 22, 29 and 43 after initial investigational product application. The investigational products were used topically during the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarchal female subjects must have a negative urine pregnancy test
* Willing to provide written informed consent/assent
* Diagnosed as having mild to moderate Atopic Dermatitis (AD)
* Willing to stop all moisturizers and/or other skin barrier cream or emulsion treatments for the AD condition during the test period and replace with the investigational product assigned in this trial
* Willing to replace their body wash and/or soaps with the one provided in this trial

Exclusion Criteria:

* Severe AD as determined by the Rajka-Langeland Severity Index
* AD requiring systemic, super-potent (Class I) or potent (Class II or III) topical corticosteroids. If the subject requires any of these medications as rescue therapy during the study, the subject will be discontinued from the trial
* History of allergy or hypersensitivity to the ingredients of the test devices, nuts or nut oil
* Cutaneous or systemic viral (including HIV or AIDS), mycotic or bacterial disease requiring a topical or systemic therapy
* Diabetes mellitus that cannot be controlled by diet alone (i.e., requires systemic medications for control)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide Division of Johnson & Johnson Consumer Companies, Inc.
Locations (2):
- United States (2):
  - Thomas J. Stephens & Associates, Inc, Colorado Springs, Colorado
  - Academic Dermatology Associates, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Device: Investigational Device - Apply 3 times daily (or as needed) on all body areas, including the affected areas of the body and face throughout duration of the study. Massage gently into skin.
- Atopiclair® Skin and Wound Emulsion: Atopiclair® Skin and Wound Emulsion - Apply 3 times daily (or as needed) on all body areas, including the affected areas of the body and face throughout duration of the study. Massage gently into skin.
Period: Overall Study
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Started | 41 | 41
Completed | 37 | 39
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.37 (2.90) | 5.56 (2.84) | 5.96 (2.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 28 | 46
  Male | 23 | 13 | 36
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Eczema Area and Severity Index (EASI) Score on Day 43 - Change From Baseline
Description: The surface and severity of eczema is measured using the Eczema Area and Severity Index (EASI). A regional body surface area tabulation based on severity ranging from 0 (none) to 3 (severe), and severity of signs of disease, then multiplied by body area with final possible calculation ranging from 0 (none) - 72 (severe).
Time Frame: Baseline to Day 43
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Number analyzed (Participants) | 39 | 40
units on a scale | -4.97 (0.41) | -5.01 (0.40)
Statistical Analysis 1: Comparison: Investigational Device vs Atopiclair® Skin and Wound Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.9416, Repeated measures ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment, visit number, and treatment-visit number interaction term as factors, with baseline score and age as covariates; Estimated Mean Difference = 0.04, 95% CI 2-sided [-1.09 to 1.17]

2. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 15 - Change From Baseline
Description: as for outcome 1
Time Frame: Baseline to Day 15
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Number analyzed (Participants) | 35 | 41
units on a scale | -3.79 (0.41) | -4.14 (0.40)
Statistical Analysis 1: Comparison: Investigational Device vs Atopiclair® Skin and Wound Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.5431, Repeated measures ANCOVA — The significance level threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Mean Difference = 0.35, 95% CI 2-sided [-0.78 to 1.48]

3. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 43 - Change From Baseline
Description: The signs and symptoms of eczema are measured using the Investigator's Global Atopic Dermatitis Assessment (IGADA), with possible values of clear (0), almost clear (1), mild (2), moderate (3), severe (4), or very severe (5).
Time Frame: Baseline to Day 43
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Number analyzed (Participants) | 41 | 41
units on a scale | 0.78 (0.15) | 0.73 (0.15)
Statistical Analysis 1: Comparison: Investigational Device vs Atopiclair® Skin and Wound Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.788, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment as a factor, baseline score as covariate; Estimated Mean Difference = -0.06, 95% CI 2-sided [-0.47 to 0.36]

4. Secondary Outcome: Itch Score on Day 43 - Change From Baseline
Description: The subject's and/or caregiver's assessment of itch was measured on a 10-cm visual analog scale (VAS) in which 0 cm represented no itch and 10 cm represented worst itch imaginable.
Time Frame: Baseline to Day 43
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Number analyzed (Participants) | 37 | 36
units on a scale | -3.26 (0.33) | -3.29 (0.33)
Statistical Analysis 1: Comparison: Investigational Device vs Atopiclair® Skin and Wound Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.9508, Repeated measures ANCOVA — The significance threshold level was 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]; Estimated Mean Difference = 0.03, 95% CI 2-sided [-0.90 to 0.96]

ADVERSE EVENTS:
Time Frame: Day 43, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 8 (Day 43). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Investigational Device | Atopiclair® Skin and Wound Emulsion
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 15/41 | 12/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Device (N=41) | Atopiclair® Skin and Wound Emulsion (N=41)
Application Site Irritation (General disorders) | 7 | 11
Application Site Pain (General disorders) | 9 | 7
Gastroenteritis (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed not to publish the study results without prior sponsor approval.